CLINICAL TRIAL: NCT03469921
Title: Unicentric Retrospective Analysis of a Cohort of 602 Young Adult and Adolescent Patients (AJA), Aged 15 to 30 Years, With Haematological Malignancies, and Managed Between 2000 and 2016
Acronym: HEMAJA
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: HEMAJA-IPC 2017-045
Record Dates: First submitted 2018-03-05; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Malignant Haemopathies; Acute Leukemia; Non-hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Malignant haemopathies; Acute Leukemia; Non-hodgkin Lymphoma; Hodgkin Lymphoma; Young adults; Adolescent
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- 15-17 years old: 15-17 years old
  Interventions: Drug: administered therapeutic regimens
- 18-25 years old: 18-25 years old
  Interventions: Drug: administered therapeutic regimens
- 26-30 years old: 26-30 years old
  Interventions: Drug: administered therapeutic regimens
- acute leukemia: acute leukemia
  Interventions: Drug: administered therapeutic regimens
- non-Hodgkin's lymphoma: non-Hodgkin's lymphoma
  Interventions: Drug: administered therapeutic regimens
- Hodgkin lymphoma: Hodgkin lymphoma
  Interventions: Drug: administered therapeutic regimens
- pediatric therapeutic regimen administered: pediatric therapeutic regimen administered
  Interventions: Drug: administered therapeutic regimens
- adult therapeutic regimen administered: adult therapeutic regimen administered
  Interventions: Drug: administered therapeutic regimens
- patients included in clinical trials: patients included in clinical trials
  Interventions: Drug: administered therapeutic regimens
- patients not included in clinical trials: patients not included in clinical trials
  Interventions: Drug: administered therapeutic regimens

INTERVENTIONS:
Drug: administered therapeutic regimens — administered therapeutic regimens

SUMMARY:
Unicentric retrospective analysis of a cohort of 602 young adult and adolescent patients, aged 15 to 30 years, with haematological malignancies, and managed between 2000 and 2016

DETAILED DESCRIPTION:
The therapeutic results (response and survival) of young adult and adolescent patients with hematological malignancies are generally lower than those usually observed in adults over the age of 30, with equivalent treatment, particularly in lymphomatous pathology.The overall analysis of this large cohort of patients in its entirety, then by age groups (15-17 years, 18-25 years, 26-30 years) and pathology aims to describe the future of patients and patients. compare them to the results of the literature observed in this age group, and according to the therapeutic regimens administered (pediatric regimen or adult regimen).

ELIGIBILITY:
Inclusion Criteria:

* Malignant hemopathies (acute leukemia, non-Hodgkin's lymphoma, Hodgkin's lymphoma) in primary care between 2000 and 2016.

Exclusion Criteria:

* Not applicable

Ages: 15 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: cohort of young adult patients and adolescents aged 15 to 30, carriers of hematological malignancies, and supported between 2000 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Global Survival | 15 years
  delay between the date of diagnosis and the date of the latest news
Survival without event | 15 years
  delay between the date of diagnosis and an event (relapse, death, lost of follow-up)
Progression-free survival | 15 years
  defined as the delay between the date of diagnosis and the date of relapse or death.

SECONDARY OUTCOMES:
Epidemiological distribution by pathology compared to the adult population over 30 years | 1 day
  Epidemiological distribution by pathology compared to the adult population over 30 years
Descriptive analysis of the characteristics of the disease at diagnosis by pathology | 15 years
  Descriptive analysis of the characteristics of the disease at diagnosis by pathology
Descriptive analysis of treatments by pathology | 15 years
  Descriptive analysis of treatments by pathology
Overall survival (OS) of patients included in clinical trials compared to patients not included for the overall cohort and pathology | 15 years
  Overall survival (OS) of patients included in clinical trials compared to patients not included for the overall cohort and pathology
Event-free survival (EFS) of patients included in clinical trials compared to patients not included for the overall cohort and pathology | 15 years
  Event-free survival (EFS) of patients included in clinical trials compared to patients not included for the overall cohort and pathology
Progression-free survival (PFS) of patients included in clinical trials compared to patients not included for the overall cohort and pathology | 15 years
  Progression-free survival (PFS) of patients included in clinical trials compared to patients not included for the overall cohort and pathology
Long-term toxicity analysis (second cancers, fertility) for the global cohort and pathology. | 15 years
  Long-term toxicity analysis (second cancers, fertility) for the global cohort and pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Diane COSO, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No